CLINICAL TRIAL: NCT01939535
Title: Prospective Evaluation of the Value of Magnetic Resonance Imaging as a One-stop-shop for Preoperative Stratification of Patients With Complexe Endometriosis - Imaging Deep Endometriosis Assessment Versus Laparoscopy.
Brief Title: Preoperative Staging of Endometriosis With MRI
Acronym: IDEAL
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S54441
Record Dates: First submitted 2013-06-27; First posted 2013-09-11 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2016-11

CONDITIONS: Endometriosis
Keywords: Endometriosis; Magnetic resonance imaging
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with endometriosis: Women with endometriosis with the intention of surgery - no intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Evaluation of an imaging technique ic MRI

SUMMARY:
The purpose of the study is to evaluate the value of MRI in preoperative stratification of endometriosis patients needing surgical approach by gynaecologists only or multidisciplinary approach by gynaecologists, urologists or/and abdominal surgeons.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the value of MRI in preoperative stratification of endometriosis patients needing either a surgical approach by gynaecologists only or multidisciplinary approach by gynaecologists, urologists or/and abdominal surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Women with strong suspicion of deep infiltrating endometriosis, with already planned surgery

Exclusion Criteria:

* Contra-indications for MRI; claustrophobic patients; patients in bad condition; pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with endometriosis in a tertiary referral centre
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Odds of changed surgical approach in deep endometriosis based on preoperative MRI findings. | All the imaging findings will be checked during a laparoscopy the latest 80 weeks after the imaging examinations.
  All endometriosis lesions found on MRI will be checked during laparoscopy in order to determine how the MRI findings might have changed the decision to do a surgical approach by gynaecologists only or multidisciplinary approach by gynaecologists, urologists or/and abdominal surgeons, and this compared to the conventional preoperative imaging approach (double contrast barium enema, intravenous urography and ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Bielen, PhD, Principal Investigator — University Hospitals KULeuven; Elvier Mussen, MD, Principal Investigator — University Hospitals KULeuven; Carla Tomassetti, MD, Principal Investigator — University Hospitals KULeuven; Christel Meuleman, PhD, Principal Investigator — University Hospitals KULeuven
Locations (1):
- University Hospitals KULeuven, Leuven, Belgium